CLINICAL TRIAL: NCT06511687
Title: Effectiveness And Impact of Nirsevimab In A Nationwide Immunization Program During The 2024 Winter Campaign In Chile (Nirse-CL)
Brief Title: Effectiveness And Impact Of Nirsevimab In Chile (NIRSE-CL)
Status: Recruiting | Type: Observational
Sponsor: Instituto Sistemas Complejos de Ingeniería (Other)
Responsible Party: Sponsor
Other Study IDs: ISCI00000001
Record Dates: First submitted 2024-07-09; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: RSV
Keywords: RSV; Nirsevimab
MeSH Terms: interventions — nirsevimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Newborns: Subjects born between April 1st, and September 31st in 2024
  Interventions: Biological: Nirsevimab
- Catch-up: Subjects born between October 1st of 2023 and March 31st of 2024
  Interventions: Biological: Nirsevimab
- High-risk: High-Risk Cohort: Infants born with 29 weeks of gestational age (wga) or less who were born within nine months of the beginning of the RSV season; those born with Bronchopulmonary Dysplasia (BPD), 32 or less wga and/or a birth weight less than 1·5 kgs born within one year of the beginning of the RSV season, and newborns 34 or less wga and/or weight less than 2·5 kgs born during the RSV season.
  Interventions: Biological: Nirsevimab

INTERVENTIONS:
Biological: Nirsevimab — Nirsevimab will be administered in a single dose at birth for newborn cohort and at the beginning of the campaign for the other cohorts under study
  Other Names: Beyfortus

SUMMARY:
The Nirse-CL study is a collaborative effort between the Ministry of Health of Chile, Instituto Sistemas Complejos de Ingeniería (ISCI), and the Faculty of Medicine of the University of Chile. The primary aim is to determine the effectiveness of the monoclonal antibody nirsevimab in preventing RSV infection in infants based on the integrated analysis of several national databases before, during, and after the implementation of a universal immunization program. The impact of the program on RSV-related health outcomes will also be determined.

DETAILED DESCRIPTION:
The primary aim of NirseCL is to evaluate the effectiveness of nirsevimab against Respiratory Syncytial Virus (RSV) in infants during the 2024 RSV season in Chile. The secondary objective is to determine the impact on RSV-related health outcomes at a national level.

The target population to receive nirsevimab is approximately 160,000 subjects, including the entire newborn cohort born during the autumn-winter season, from April 1st, 2024, to September 31st, 2024, infants born from October 1st, 2023, to March 31st, 2024, which are 6 to 1 month old at the time of immunization in April-June, and the high-risk group defined as infants born with 29 weeks of gestational age (wga) or less who were born within nine months of the beginning of the RSV season; those born with Bronchopulmonary Dysplasia (BPD), 32 or less wga and/or a birth weight less than 1·5 kgs born within one year of the beginning of the RSV season, and newborns 34 or less wga and/or weight less than 2·5 kgs born during the RSV season.

Nirsevimab will be administered as part of Chile's national immunization program, following the implementation plan designed by the Ministry of Health. The coverage with nirsevimab in the target population is expected to be high (95% for those born during the winter campaign and 80% for those born before the beginning of the autumn-winter season).

The primary outcome measure for effectiveness will be lower-tract respiratory infection hospitalizations (LRTI) attributed to RSV in the pediatric intensive care units (PICU) at a nationwide and regional level, and the secondary outcomes will be overall LRTI hospitalizations attributed to RSV, LRTI hospitalizations, and hospitalizations due to any cause. Additional outcomes might be included if enough statistical power is attained.

Effectiveness will be determined using a two-step process. First, historical data will be used to determine the set of ICD10 diagnosis codes that are attributable to RSV infection by using data from the Chilean national sentinel program and consolidated hospitalization records. Afterward, A series of complementary statistical analyses at different aggregation levels will be conducted to estimate the impact of nirsevimab on the target population. Detailed patient-level information will be used to compare LRTI hospitalizations of those receiving the immunization against those who did not, using an adjusted proportional hazard rates regression model to estimate the effectiveness of nirsevimab as a function of covariates such as wga, weight at birth, sex, nationality, maternal education, coexisting conditions, MMR vaccination (as an indicator of access to medical care), and place of birth. This method has been used to evaluate recent nationwide vaccination campaigns in Chile (Jara et al, 2021). A case-control matching approach will be used as an alternative method intended to gain statistical efficiency (Rose and van der Laan, 2009). Finally, as a robustness analysis, a synthetic control method that allows the comparison of whole time series without relying on individual-level data will be used (Bruhn et al., 2016).

ELIGIBILITY:
Inclusion Criteria:

* Subjects born between October 1st, 2023, to September 31st, 2024.
* Subjects born with 29 weeks of gestational age (wga) or less who were born between July 1st, 2023 and October 1st, 2023
* Subjects born with Bronchopulmonary Dysplasia (BPD), 32 or less wga and/or a birth weight less than 1·5 kgs born between April 1st, 2023 and October 1st, 2023.

Exclusion Criteria:

* No specific criteria has been reported

Max Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All infants born in Chile between October 1st, 2023, to September 31st, 2024 (approximately 160.000), and all high-risk infants born between July 1st, 2023, and October 1st, 2023 (approximately <1.000).
Sampling Method: Non-Probability Sample
Enrollment: 160000 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
LRTI | from April 2024 to October 2024
  Number and incidence of lower-tract respiratory infections hospitalizations (LRTI) attributed to RSV in the pediatric intensive care units (PICU) at a nationwide and regional level.

CONTACTS AND LOCATIONS:
Locations (1):
- ISCI, Santiago, Chile

REFERENCES:
- [Background] Rose S, Laan MJ. Why match? Investigating matched case-control study designs with causal effect estimation. Int J Biostat. 2009 Jan 6;5(1):Article 1. doi: 10.2202/1557-4679.1127. PMID 20231866
- [Background] Martens L, Leroy R, Jara A, Garcia-Zattera MJ, Lesaffre E, Declerck D. Variables associated with longitudinally registered plaque accumulation in a cohort of Flemish schoolchildren. Quintessence Int. 2007 Jul-Aug;38(7):555-64. PMID 17694211
- [Background] Bruhn CA, Hetterich S, Schuck-Paim C, Kurum E, Taylor RJ, Lustig R, Shapiro ED, Warren JL, Simonsen L, Weinberger DM. Estimating the population-level impact of vaccines using synthetic controls. Proc Natl Acad Sci U S A. 2017 Feb 14;114(7):1524-1529. doi: 10.1073/pnas.1612833114. Epub 2017 Feb 1. PMID 28154145
- [Background] Pearce N. Analysis of matched case-control studies. BMJ. 2016 Feb 25;352:i969. doi: 10.1136/bmj.i969. PMID 26916049
- [Derived] Torres JP, Saure D, Goic M, Thraves C, Pacheco J, Burgos J, Trigo N, Del Solar F, Neira I, Diaz G, O'Ryan M, Basso LJ. Effectiveness and impact of nirsevimab in Chile during the first season of a national immunisation strategy against RSV (NIRSE-CL): a retrospective observational study. Lancet Infect Dis. 2025 Nov;25(11):1189-1198. doi: 10.1016/S1473-3099(25)00233-6. Epub 2025 Jun 10. PMID 40513593